CLINICAL TRIAL: NCT03592303
Title: Bedside Assessment of Coagulation in Post-partum Hemorrhage by Thromboelastography (TEG ®6S)
Acronym: HPPTEG6S
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI17042J; 2017-A02347-46 (Other: ANSM)
Record Dates: First submitted 2018-04-27; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-05

CONDITIONS: Coagulation Defect; Puerperal; Post Partum Hemorrhage; Blood Protein Disorders; Pregnancy Hemorrhage
Keywords: Post-partum haemorrhage; Thromboelastography; Coagulopathy; Fibrinogenemia
MeSH Terms: conditions — Hemostatic Disorders; Postpartum Hemorrhage; Blood Protein Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Any pregnant patient with a normal pregnancy is eligible for possible participation in the study.
- PPH group: Women with PPH requiring biological evaluation of hemostasis

SUMMARY:
Postpartum hemorrhage (PPH) is one of the leading causes of maternal deaths. Its prognosis is directly influenced by the early diagnosis and treatment of the associated coagulopathy. In this context, fibrinogen concentration is the best predictor of a severe PPH. The medical interest of thromboelastography/elastometry to early detect and guide the rapid correction of coagulopathy in PPH is regularly discussed.

The principal aim of this study is to evaluate the performance of a new hemostasis point of care device (thromboelastography - TEG ®6S) for the diagnosis of coagulopathy during PPH.

A secondary aim will be to determine the normal values of TEG6S at the end of a normal pregnancy.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a complication of 5 to 10% of deliveries and is the leading cause of maternal mortality, all over the world. In France, as in other developed countries, 20% of maternal mortality is related to PPH complications with a high rate of avoidance (85%) due to inappropriate or delayed therapeutic measures). The management of PPH is based on recommendations highlighting the need for early detection and treatment of coagulopathy, which is predictive of the hemorrhage severity. The prognosis of the PPH is directly related to the rapidity of the coagulopathy treatment (30 to 60 minutes after diagnosis). Severe PPH is often associated with clotting disorders of either primary origin (disseminated intravascular coagulation) or secondary origin (coagulation factors loss due to hemorrhage). A hypofibrinogenemia < 2 g/L is the best predictor of a severe PPH with a positive predictive value of 100% . Similarly, abnormal coagulation tests appear to be predictive of the severity of the bleeding and the subsequent need for invasive procedures.

The assessment of coagulation is currently based on standard laboratory hemostasis tests, but with delayed time to obtain results, generally greater than 60 minutes. Therefore, early and fast assessment of hemostasis during PPH is essential to estimate the bleeding severity and allow early and adequate administration of pro-coagulant products, leading to an improved prognosis of PPH. The medical interest of thromboelastography (TEG) to early diagnose and guide the treatment of a coagulopathy in PPH is regularly discussed.

A previous observational study performed by our team in 2013 during PPH (95 patients and133 samples) compared the TEG 5000 parameters with the standard laboratory hemostasis tests. Our results confirm the good predictability of TEG 5000 for the early detection of a hypofibrinogenemia ≤ 2 g / l and/or thrombocytopenia ≤ 80 000 platelets / mm3 (AUC between 0.91 and 0.97). Among the biological parameters analyzed by the TEG 5000, the parameters K-MRTGG and FF-MRTGG (maximum rate of thrombus generation) were also evaluated. Their predictabilities were as good as the usual K-MA or FF-MA (comparable AUC) and were available more rapidly than usual parameters (3 ± 3 min for FF-MRTGG and 8 ± 3 min for K-MRTGG), allowing a very early evaluation of hemostasis.

The aim of this prospective observational study is therefore to evaluate the performance of a new delocalized hemostasis monitoring device (thromboelastography - TEG ®6S) for the diagnosis of coagulopathy during PPH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient with health insurance
* Group of patients during labor : any pregnant woman with a normal pregnancy in the delivery room.
* Group of patients with PPH: any woman with a normal pregnancy experiencing a PPH with blood loss greater than 500 mL and who requires a biological evaluation of haemostasis.

Exclusion Criteria:

* Coagulopathy pre-existing to pregnancy
* Medication that interferes with blood coagulation
* Hepato-cellular insufficiency
* Renal failure
* Psychiatric care patients
* Patient deprived of liberty by judicial or administrative decision
* Major patient undergoing legal protective measures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any pregnant patient with a normal pregnancy is eligible for possible participation in the study.
  Two patient groups will be included :
  * Pregnant women during labor
  * Women with PPH requiring biological evaluation of hemostasis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Performance analysis of TEG6S kaolin parameters for the diagnosis of coagulation disorders in PPH. | during the 24 hours after delivery
  The performance analysis of the parameters derived from the Kaolin test will be performed using ROC curves and a sensitivity and specificity calculation.

SECONDARY OUTCOMES:
Performance analysis of TEG6S RapidTEG parameters for the diagnosis of coagulation disorders in PPH. | during the 24 hours after delivery.
  The performance analysis of the parameters derived from the RapidTEG test will be performed using ROC curves and a sensitivity and specificity calculation.
Performance analysis of TEG6S Functional Fibrinogen parameters for the diagnosis of coagulation disorders in PPH. | during the 24 hours after delivery.
  The performance analysis of the parameters derived from Functional Fibrinogen test will be performed using ROC curves and a sensitivity and specificity calculation.
Analysis of the correlation between the parameters provided by TEG6S and standard laboratory tests. | during the 24 hours after delivery.
  Analysis of correlation between the parameters of CFF test and laboratory tests.
Analysis of the correlation between the parameters provided by TEG6S and standard laboratory tests.standard laboratory tests. | during the 24 hours after delivery.
  analysis of correlation between the parameters of CK test and laboratory tests.
Analysis of the correlation between the parameters provided by TEG6S and standard laboratory tests. | during the 24 hours after delivery.
  analysis of correlation between the parameters of CRT test and laboratory tests.
Performance of TEG6S parameters for predicting severe HPP | 24 hours after delivery.
  Blood loss will be calculated 24 hours after delivery, based on demographic data and hematocrit (Ht) values measured in the last month of pregnancy and 24 hours after delivery.
Comparison of the time taken to obtain the different TEG6S parameters versus standard biology parameters. | during 24 hours after delivery
  The time taken to obtain the TEG6S parameter CK-MA will be measured. It corresponds to the time between the start of the analysis (including the start of the test) and the time the result is provided by the TEG6S.
Comparison of the time taken to obtain the different TEG6S parameters versus standard biology parameters. | during 24 hours after delivery
  The time taken to obtain the TEG6S parameter CRT-MA will be measured. It corresponds to the time between the start of the analysis (including the start of the test) and the time the result is provided by the TEG6S.
Comparison of the time taken to obtain the different TEG6S parameters versus standard biology parameters. | during 24 hours after delivery
  The time taken to obtain the TEG6S parameter FF-MA will be measured. It corresponds to the time between the start of the analysis (including the start of the test) and the time the result is provided by the TEG6S.
Define normal reference values for TEG6S Thromboelastography in pregnant women during labor. | during 24 hours after delivery
  2.9 mL of additional blood will be collected for TEG6S analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Agnès Rigouzzo, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Trousseau, Paris, France